CLINICAL TRIAL: NCT04452266
Title: Predictive Factor Study of the Occurrence of Endometrial Cancer in Patients With Lynch Syndrome: Study Conducted in the Hauts-de-France
Brief Title: Predictive Factor Study of the Occurrence of Endometrial Cancer in Patients With Lynch Syndrome
Acronym: PrediLynch
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_07; 2020-A00843-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Lynch Syndrome
Keywords: lynch syndrome; endometrial cancer
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Women with Lynch Syndrome and endometrial Cancer matched on age of endometrial cancer diagnosis
  Interventions: Other: questionnaire assesment
- control group: Women with Lynch Syndrome, without Cancer at Lynch Syndrome Diagnostic matched on their age at Lynch Diagnostic
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — Each patient will to answer questions about their medical history.

SUMMARY:
Lynch Syndrome increases Endometrial Cancer Occurrence in women due to failure in MisMatch Repair System. Lifetime Cumulative risk of developing endometrial Cancer is approximatively 40% in women with Lynch Syndrome.

Endometrial cancer is the third women cancer in France. Many risk factors are known in general population. Lots of factors are related to over exposure to estrogen.

Data about influence of general risk factors in Women with Lynch Syndrome are poor. Recently, a cohort study appears to have shown a significant decrease in the risk of endometrial cancer with multiparity, the use of hormonal contraception and late menopause in Lynch women. The impact of weight and certain metabolic parameters on the occurrence of endometrial cancers remains poorly known to this day.

ELIGIBILITY:
Inclusion Criteria:

* Lynch Syndrome Diagnosis at University Hospital
* Alive at study time
* Age over 30 at endometrial cancer or Lynch Syndrome Diagnosis

Case group :

- No cancer before endometrial cancer diagnosis

Control group :

* No endometrial cancer developped
* Free cancer women at Lynch Syndrome diagnosis

Exclusion Criteria:

* Refusing to participate
* Poor understanding of the French language
* Other cancer diagnosed before endometrial cancer
* Hysterectomy before lynch diagnosis for free cancer women

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — woman
Study Population: Women included are all carriers of Lynch syndrome, already diagnosed by genetic analysis in the Molecular Biology Laboratory of the CHU de Lille and whose analysis was transmitted during a consultation at the Guy Fontaine Genetics Clinic during the period from 01/01/1998 to 30/11/2019 at the CHU de Lille or in advanced consultations in the regions.The database PROGENY will be use to extract population corresponding to the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Correlation between endometrial cancer and predictif factors | Baseline
  Endometrial cancer (yes/no) and explicative variable: Diabetes before endometrial cancer or Lynch syndrome diagnosis; Smoking ; Maximal Weight ; Age at menarche; Parity ; Age at first birth ; Contraceptive use.

SECONDARY OUTCOMES:
Correlation between endometrial cancer and predictif factors in post menopausal woman | Baseline
  Endometrial cancer (yes/no) and explicative variable: Menopause age; Hormonal menopause treatment

CONTACTS AND LOCATIONS:
Overall Officials: Solveig MENU-HESPEL, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, Lille, France

IPD SHARING:
Plan to Share IPD: No